CLINICAL TRIAL: NCT06016062
Title: A Multi-center Phase I/II Trial to Evaluate the Efficacy and Safety of RC148 As a Single Agent and Combination Therapy in Patients with Locally Advanced Unresectable or Metastatic Malignant Solid Tumors
Brief Title: A Study of RC148 As a Single Agent and Combination Therapy in Patients with Locally Advanced Unresectable or Metastatic Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC148-C001
Record Dates: First submitted 2023-08-18; First posted 2023-08-29 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Phase1-RC148 monotherapy (Experimental): Participants will be allocated to one of the following dose groups:1.0, 3.0, 10.0, 20.0, and 30.0mg/kg, and receive a treatment of RC148 followed by 28 days of dose limited toxicity (DLT) observation period.
  Interventions: Drug: RC148 Monotherapy
- Phase2-Arm1 (NSCLC): RC148+docetaxel (Experimental): RC148+docetaxel Combination Therapy： Participants receive RC148 (10mg/kg or 20mg/kg Q3W) in combination with docetaxel (75mg/m^2 Q3W).
  Interventions: Drug: RC148+docetaxel Combination Therapy
- Phase2-Arm 2 (Cervical): RC148+RC48 (Experimental): RC148+RC48 Combination Therapy:
  Participants receive RC148 (20mg/kg Q2W) in combination with RC48 (2.0mg/kg Q2W).
  Interventions: Drug: RC148+RC48 Combination Therapy
- Phase2-Arm 3 (Gastric cancer) : RC148+RC48 (Experimental): RC148+RC48 Combination Therapy: Participants receive RC148 (20mg/kg Q2W) in combination with RC48 (2.0mg/kg Q2W).
  Interventions: Drug: RC148+RC48 Combination Therapy
- Phase2-Arm 4 (Lung Adenocarcinoma): RC148+RC88 (Experimental): RC148+RC88 Combination Therapy: Participants receive RC148 (20mg/kg Q3W) in combination with RC88 (2.0mg/kg Q3W).
  Interventions: Drug: RC148+RC88 Combination Therapy
- Phase2-Arm 5 (Platinum-resistant Ovarian cancer) : RC148/Bevacizumab+RC88 (Experimental): RC148+RC88 Combination Therapy: Participants receive RC148 (20mg/kg Q3W) in combination with RC88 (2.0mg/kg Q3W).
  Bevacizumab+RC88 Combination Therapy: Participants receive Bevacizumab (15mg/kg Q3W) in combination with RC88 (2.0mg/kg Q3W).
  Interventions: Drug: RC148/Bevacizumab+RC88 Combination Therapy
- Phase2-Arm 6 (Platinum-sensitive Ovarian cancer): RC148+RC88 (Experimental): RC148+RC88 Combination Therapy: Participants receive RC148 (20mg/kg Q3W) in combination with RC88 (2.0mg/kg Q3W).
  Interventions: Drug: RC148+RC88 Combination Therapy
- Phase2-Arm 7 (MSLN-expressing Cervical cancer): RC148+RC88 (Experimental): RC148+RC88 Combination Therapy: Participants receive RC148 (20mg/kg Q3W) in combination with RC88 (2.0mg/kg Q3W).
  Interventions: Drug: RC148+RC88 Combination Therapy

INTERVENTIONS:
Drug: RC148 Monotherapy — RC148 injection will be administered as an intravenous (IV) infusion on Day 1 of each 3-week cycle
  Other Names: RC148 for injection
  Arms: Phase1-RC148 monotherapy
Drug: RC148+docetaxel Combination Therapy — RC148 injection will be administered as an intravenous (IV) infusion on Day 1 of each 3-week cycle； Docetaxel will be administered as an IV infusion on Day 1 of each 3-week cycle.
  Arms: Phase2-Arm1 (NSCLC): RC148+docetaxel
Drug: RC148+RC48 Combination Therapy — RC148 injection will be administered as an intravenous (IV) infusion on Day 1 of each 2-week cycle； RC48 will be administered as an IV infusion on Day 1 of each 2-week cycle.
  Arms: Phase2-Arm 2 (Cervical): RC148+RC48; Phase2-Arm 3 (Gastric cancer) : RC148+RC48
Drug: RC148+RC88 Combination Therapy — RC148 injection will be administered as an intravenous (IV) infusion on Day 1 of each 3-week cycle； RC88 will be administered as an IV infusion on Day 1 of each 3-week cycle.
  Arms: Phase2-Arm 4 (Lung Adenocarcinoma): RC148+RC88; Phase2-Arm 6 (Platinum-sensitive Ovarian cancer): RC148+RC88; Phase2-Arm 7 (MSLN-expressing Cervical cancer): RC148+RC88
Drug: RC148/Bevacizumab+RC88 Combination Therapy — RC148 injection will be administered as an intravenous (IV) infusion on Day 1 of each 3-week cycle; RC88 will be administered as an IV infusion on Day 1 of each 3-week cycle; Bevacizumab will be administered as an IV infusion on Day 1 of each 3-week cycle
  Arms: Phase2-Arm 5 (Platinum-resistant Ovarian cancer) : RC148/Bevacizumab+RC88

SUMMARY:
The primary objective of Phase I of this trial is to evaluate the safety, tolerability, maximum tolerated dose (MTD)/maximum administered dose (MAD) of RC148 in patients with locally advanced unresectable or metastatic solid tumors to determine the recommended Phase II dose (RP2D), and the secondary objective is to evaluate the PK and PD characteristics, immunogenicity and preliminary clinical efficacy of RC148. Phase II will primarily evaluate the efficacy of the RC148 combination regimen, and secondarily will assess safety and tolerability, PK characteristics, and immunogenicity. During the trial, investigators will also evaluate the potential correlation of biomarkers with efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to participate in the study voluntarily and willing to provide written informed consent.
2. male or female ≥18 years (phase Ⅰ), 18 to 75 years old (Including 18 and 75 years, phase Ⅱ).
3. Must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
4. Projected life expectancy of at least 12 weeks.
5. At least one measurable target lesion based on imaging according to RECIST v1.1 criteria (For patients who have received prior radiotherapy, radiotherapy-treated lesions may be considered as target lesions if the lesion is measurable according to RECIST v1.1 criteria and there is evidence of significant progression after radiotherapy.);
6. Requirements for inclusion of subjects at different stages:

   Phase I (RC148 monotherapy): Patients with locally advanced unresectable or metastatic malignant solid tumors whose disease has progressed with standard therapy, or who are unable to tolerate standard therapy, or in whom the subject refuses standard therapy;

   Phase II (Combination Therapies):

   Cohort 1 (non-small cell lung cancer): Patients with locally advanced unresectable or metastatic malignant solid tumors with disease progression on standard therapy, or intolerance of standard therapy, or refusal of standard therapy.

   Cohort 2 (HER2-expressing cervical cancer): Subjects with advanced non-small cell lung cancer diagnosed by histological or cytological examination, locally advanced or metastatic, with AGA- confirmed by prior genetic testing, who have received a PD-1/PD-L1 inhibitor and platinum-based chemotherapy as a first or second-line advanced treatment, and who have not received docetaxel chemotherapy.

   Cohort 3 (HER2 expressing gastric cancer): Histologically and/or cytologically confirmed locally advanced or metastatic gastric adenocarcinoma (including gastroesophageal junction adenocarcinoma) with HER2 expression (IHC ≥1+). Subjects who have progressed or are intolerant to standard first-line therapy only (PD-1/PD-L1 inhibitor + platinum-containing chemotherapy ± trastuzumab, and not including paclitaxel). Disease progression during neoadjuvant therapy and within 6 months of the end of adjuvant therapy will also be considered a failure of first-line therapy.

   Cohort 4 (MSLN-expressing lung adenocarcinoma): Histologically or cytologically confirmed lung adenocarcinoma without other pathologic components; driver gene negative, MSLN-expressing (IHC ≥1+) advanced lung adenocarcinoma subjects who have received PD-1/PD-L1 inhibitor and platinum-based chemotherapy (combination or sequential) and have not received paclitaxel-based chemotherapy.

   Cohort 5 (platinum-resistant ovarian, fallopian tube, or primary peritoneal cancer): pathologic type needs to be high-grade serous ovarian cancer; Subjects who have progressed on prior 1-4 lines of antitumor therapies; Definition of platinum-resistance: 1) Patients who have received 1 line of platinum-based therapy must have received at least 4 cycles of platinum, must have had a response (CR or PR), and then progressed between >3 months and ≤6 months after the date of the last platinum; 2) Patients who have received 2 or 3 lines of platinum-based therapies must have received at least 4 cycles of platinum and have progressed on or within 6 months after the last dose of platinum.

   Cohort 6 (platinum-sensitive ovarian, fallopian tube, or primary peritoneal cancer): Pathological type needs to be high-grade serous EOC; Subjects who have received 1-4 lines of prior antitumor therapies were included.

   Cohort 7 (MSLN-expressing cervical cancer): Subjects with recurrent or metastatic cervical cancer expressing mesothelin (MSLN) (IHC ≥1+) that is histologically confirmed, ineligible for surgery or radiotherapy, and has progressed after at least 1L of platinum-based chemotherapy.
7. Participants agree to provide pre-treatment archived/biopsied tumor samples for biomarker-related testing such as retrospective programmed cell death protein 1 (PD-L1) expression levels. Biopsies will be considered at screening only if archived samples are not available. Fresh tumor biopsies will not be considered if significant risk procedures are required per the discretion of the Investigator.
8. Adequate bone marrow, liver, and renal function defined as:

   No platelet or red blood cell transfusion within 14 days prior to performing routine blood tests, no correction with thrombopoietin (TPO), erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF), or interleukin-11 (IL-11), absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L, platelets ≥ 100 × 10^9/L, and Hemoglobin ≥ 90g/L.

   Serum total bilirubin ≤1.5 × upper limit of normal (ULN), ALT, AST ≤2.5 × ULN (≤5 × ULN in case of known liver metastases), albumin ≥30 g/L International Normalized Ratio (INR) ≤1.5×ULN, Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN.

   Serum creatinine ≤ 1.5 x ULN. Urinalysis results for urinary protein <++.
9. For subjects in Cohort 1 (Non-Small Cell Lung Cancer) and Cohort 4 (Lung Adenocarcinoma) of the Phase II Combined Protocol, pulse oximetry (O2 saturation) measured under unoxygenated conditions was required to be >92%.
10. Cardiac function: left ventricular ejection fraction ≥50%.
11. Male or female subjects with fertility must agree to take effective contraceptive measures during the study period and within 6 months after the end of the last medication, such as double-barrier contraceptive methods, condoms, oral or injectable contraceptives, intrauterine contraceptive device.

Exclusion Criteria:

1. Pregnant or lactating.
2. Cohort 1 in Phase II, patients with histologically or cytologically confirmed non-small cell lung cancer, other than squamous lung cancer and lung adenocarcinoma, (including subjects with squamous or adenocarcinoma in combination with other pathologic types of non-small cell lung cancer;) prior treatment with docetaxel, or an antitumor agent that targets VEGF/VEGFR; and treatment with at least 2 cycles of an immune checkpoint inhibitor, with a best response of PD, or best response of CR/PR/SD with disease progression within 6 months of first dose.
3. Cohorts 4-7 in Phase II, patients with ocular corneal conditions at screening such as congenital corneal dystrophy, meibomian gland dysfunction (MGD), viral keratitis (dendritic, map-like, corneal stromal keratitis), uveitis, corneal endothelial decompensation, glaucoma, iridocorneal endothelial syndrome (ICE).
4. Subjects with active hepatitis B or C; human immunodeficiency virus (HIV)-positive subjects.
5. Those who have received a live vaccine within 28 days prior to the first RC148 administration or who plan to receive any live vaccine during the study period.
6. Participant with a history of other acquired/congenital immunodeficiency diseases or organ transplantation.
7. Active autoimmune disease requiring systemic therapy, such as systemic lupus erythematosus, psoriasis requiring systemic therapy, or rheumatoid arthritis, within the past 2 years; however, alternative therapies are not considered systemic therapies and are permitted for use and enrollment.
8. Subject has received an immune checkpoint inhibitor (anti-PD-1/PD-L1/CTLA-4 antibody) or other immune checkpoint inhibitor therapy within 28 days prior to initiation of treatment with the study drug or has experienced permanent discontinuation of immunotherapy due to toxicity of immune checkpoint inhibitor therapy prior to receiving administration of the study drug.
9. Subjects who have participated in a clinical trial of another drug and received the test drug within 4 weeks prior to the first dose of RC148.
10. Prior concomitant treatment with antitumor agents targeting VEGF/VEGFR and PD-1/PD-L1 (except for subjects with cervical cancer). For cohorts 2-3 in Part 2, subjects with prior antibody-drug conjugates treatment. For cohorts 4-7 in Part 2, subjects with prior antibody-drug conjugates and MSLN-targeting drugs.
11. Known hypersensitivity or delayed hypersensitivity to certain components of the study drug or to similar drugs.
12. Participant who are under the treatment of anticoagulant drugs. Participants using prophylactic doses of heparin are eligible in the study.
13. Subject received last systemic antitumor therapy, including surgery, chemotherapy, radiotherapy, and biologic therapy within 4 weeks prior to the first study drug administration; received small molecule tyrosine kinase inhibitor therapy or immunotherapy within 2 weeks prior to the first drug administration; or received herbal therapy for antitumor indications within 1 week prior to the first drug administration or received bone/other solitary metastases within 2 weeks prior to the first study drug administration Palliative radiotherapy.
14. Previous adverse reactions resulting from previous anti-tumour therapies, which have not returned to Grade 1 according to NCI-CTCAE v5.0 at screening.
15. Presence of grade ≥2 sensory or motor neuropathy.
16. Presence of third interstitial fluid with clinical symptoms or requiring intervention.
17. Active infection of clinical significance judged by the investigator.
18. Active gastrointestinal bleeding, history of hemoptysis, peptic ulcer, or a hemorrhagic event with NCI CTCAE (V5.0) ≥ grade 2 within 4 weeks prior to screening; or the presence of severe esophagogastric varices, nosebleeds; and in the case of subjects with gastric cancer, a tumor lesion with a tendency to bleed.
19. Presence of systemic diseases that, in the judgment of the investigator, are not under stable control, including diabetes mellitus, hypertension, cirrhosis of the liver, etc.
20. Those with previous and current clinical manifestations or high risk factors for interstitial lung disease (ILD), drug-associated pneumonia, radiation pneumonitis, severely impaired lung function, or suspected interstitial lung disease.
21. Clinically relevant pyelonephrosis that cannot be reduced by ureteral stenting or percutaneous drainage.
22. History of gastrointestinal perforation and/or fistula, gastrointestinal obstruction, inflammatory bowel disease, or bowel resection within the past 6 months.
23. Screening QTc interval >450 ms (males), QTc interval >470 ms (females); previous family or personal history of long/short QT interval syndrome; history of ventricular arrhythmia considered clinically significant by the investigator or currently receiving antiarrhythmic medications or implantation of an arrhythmia defibrillation device.
24. Experienced an arterial/venous thromboembolic event such as cerebrovascular accident, deep vein thrombosis, pulmonary embolism, cerebral infarction, or experienced a history of hypertensive crisis or hypertensive encephalopathy within 6 months prior to initiation of study treatment.
25. History of myocardial infarction, severe or unstable angina pectoris, coronary or peripheral artery bypass graft or vascular disease, New York Heart Association (NYHA) grade ≥3 heart failure within 6 months prior to screening; history of fulminant, acute, chronic relapsing, or persistent myocarditis, pericarditis, or epicarditis from any cause within 1 year prior to screening.
26. Subjects on systemic therapy with corticosteroids (daily prednisone ≥10 mg/day or equivalent dose of drug) or other immunosuppressive medications within 2 weeks of first study administration.
27. Subjects with the presence of brain metastases who have been previously treated for brain metastases may be considered for enrollment (exclusion of brain metastases from gastric cancer): provided that the disease is stable, no disease progression has occurred as determined by imaging within 4 weeks prior to dosing, and all neurological symptoms have returned to baseline levels, and that the use of radiation, surgical, or steroid therapy has been discontinued for at least 28 days prior to the first dose of the drug; in the case of carcinomatous meningeal metastases, regardless of their clinical stabilization of symptoms, should be excluded.
28. Major surgery or intervention with incomplete recovery (except tumor biopsy or puncture) within 4 weeks prior to the first dose of study drug; or gross needle aspiration biopsy or other minor surgery, excluding placement of vascular infusion devices, within 7 days prior to initiation of study drug therapy.
29. Screening imaging showing tumor invasion of large blood vessels or imaging evidence of tumor invasion of vital organs or risk of developing a fistula; or imaging evidence of tumor encircling a large blood vessel or entry into the study causing a risk of hemorrhage.
30. Other malignancies were present within 5 years before the initiation of study administration, except for malignancies that would be expected to be cured with treatment.
31. Previous or current uncontrollable mental illness.
32. Subjects with poor compliance who were not expected to cooperate in completing trial procedures.
33. Any other disease, metabolic abnormality, physical examination abnormality, or laboratory test abnormality that, in the judgment of the Investigator, gives reason to suspect that the subject has a disease or condition that makes the subject unsuitable for the use of the investigational drug, or that would interfere with the interpretation of the results of the study, or that would place the subject at high risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase I：Maximum tolerated dose (MTD)/Maximum administered dose (MAD) | Subjects will be treated and observed for DLT through the end of the first cycle (Days 1-28)
  MTD/MAD based on number of Dose limiting toxicity (DLT)
Phase I：DLT | 28 days after first treatment
  In the DLT evaluation window (observation period 1-28 days after the first administration), according to the NCI-CTCAE v5.0 grading standard, the investigator or the sponsor believes that toxic reaction which are reasonably related to RC148 treatment
Phase I：The incidence and severity of adverse events (AE) | From the day of ICF sign to 28/90 days after the day of the last treatment
  Adverse events were assessed by investigator(s) according to NCI-CTCAE v5.0
Phase I：Recommended Phase 2 dose (RP2D) | 28 days or 1cycle
  The RP2D may be selected as 1 dose level lower than the MTD and will be determined in discussion with the safety monitoring committee based on all available data
Phase II: ORR, DCR, DoR, PFS based on RECIST v1.1 investigator assessment; | 15 months

SECONDARY OUTCOMES:
Phase I：Overall Response Rate (ORR) | 15 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)
Phase I：DCR | 15 months
  Disease Control Rate was defined as the percentage of participants with a CR or PR or stable disease (SD)
Phase I：DOR | 15 months
  Duration of response is the length of time that a tumor continues to respond to treatment without the cancer growing or spreading
Phase I：PFS | 15 months
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Phase I：Pharmacodynamic characterization of RC148 | 15 months
  PD-1 receptor occupancy in circulating T cells
Phase I：Pharmacodynamic characterization of RC148 | 15 months
  Plasma free VEGF, total VEGF levels
Phase I/II：Pharmacokinetics (PK) parameter | 15 months
Phase I/II：ADA incidence rate | 15 months
Phase II：- Incidence and severity of adverse events/serious adverse events (graded based on NCI CTCAE V5.0); | 15 months
Phase II：- Vital signs, physical examination, ECOG physical status score, 12-lead electrocardiogram, laboratory tests; | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Fang, Ph.D, Study Director — RemeGen Co., Ltd.
Locations (31):
- China (31):
  - Anhui Provincial Hospital, Anhui
  - Beijing Tiantan Hospital, Capital Medical University, Beijing
  - Beijing University Cancer Hospital, Beijing
  - The Fifth Medical Center of Chinese PLA General Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - Hunan Second People's Hospital, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The Second Affiliated Hospital of Guilin Medical University, Guilin
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jinan Central Hospital, Jinan
  - Qilu Hospital of shangdong university, Jinan
  - Shandong Cancer Hospital, Jinan
  - Meizhou People's Hospital, Meizhou
  - Guangxi Medical University Cancer Hospital & Guangxi Cancer Institute, Nanning
  - Nanyang City Center Hospital, Nanyang
  - Nanyang Second General Hospital, Nanyang
  - Shanghai Pulmonology Hospital, Shanghai
  - Liaoning Cancer Hospital & Institute, Shenyang
  - Shengjing Hospital of China Medical University, Shenyang
  - Shanxi Provincial Tumor Hospital, Taiyuan
  - Tongji Hospital, Tongji Medical College of HUST, China, Wuhan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, China, Wuhan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Yunnan Cancer Hospital, Yunnan
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No